CLINICAL TRIAL: NCT02473939
Title: A Randomised, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of VR942 in Healthy Subjects and Repeated Doses in Mild Asthmatics
Brief Title: An Evaluation of VR942 in Healthy Volunteers and Patients With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vectura Limited (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR942/1/001
Record Dates: First submitted 2015-05-29; First posted 2015-06-17 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- VR942 Dose 1 (Experimental): VR942 Dose 1
  Interventions: Drug: VR942 delivered via a Vectura Dry Powder Inhaler; Drug: Placebo delivered via a Vectura Dry Powder Inhaler
- VR942 Dose 2 (Experimental): VR942 Dose 2
  Interventions: Drug: VR942 delivered via a Vectura Dry Powder Inhaler; Drug: Placebo delivered via a Vectura Dry Powder Inhaler
- VR942 Dose 3 (Experimental): VR942 Dose 3
  Interventions: Drug: VR942 delivered via a Vectura Dry Powder Inhaler; Drug: Placebo delivered via a Vectura Dry Powder Inhaler
- VR942 Dose 4 (Experimental): VR942 Dose 4
  Interventions: Drug: VR942 delivered via a Vectura Dry Powder Inhaler; Drug: Placebo delivered via a Vectura Dry Powder Inhaler
- VR942 Dose 5 (Experimental): VR942 Dose 5
  Interventions: Drug: VR942 delivered via a Vectura Dry Powder Inhaler; Drug: Placebo delivered via a Vectura Dry Powder Inhaler

INTERVENTIONS:
Drug: VR942 delivered via a Vectura Dry Powder Inhaler
Drug: Placebo delivered via a Vectura Dry Powder Inhaler

SUMMARY:
The purpose of the study is to Evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of single inhaled doses of VR942 in healthy subjects (part 1) and repeated doses in mild asthmatics (part 2).

ELIGIBILITY:
Inclusion Criteria for Part I & 2:

* Male or female subject.
* Female subjects of non-childbearing potential
* Weigh at least 50 kg, and body mass index 18.0-31.0
* Peak inspiratory flow (PIF) of at least 60 L/min for at least 2 sec
* Forced expiratory volume in 1 sec (FEV1)/forced vital capacity (FVC) ratio of at least 0.7 at the screening visit
* Willingness to give written consent to participate after reading the information and consent form
* Willingness to give written consent to have data entered into The Over volunteering Prevention System.
* Additional inclusion criteria for Part 1:
* Healthy subjects with FEV1 and FVC of at least 80% of the predicted value at the screening visit
* Additional inclusion criteria for Part 2:
* Patients with documented clinical history of mild bronchial asthma (mild as defined by the GINA guidelines1) for at least 6 months before the screening visit
* Patient FEV1 and FVC of at least 70% of the predicted value at the screening visit

Exclusion Criteria for Part 1 & 2:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the subject's participation in the trial or make it unnecessarily hazardous (excluding mild asthma in Part 2)
* Impaired endocrine, thyroid, hepatic, respiratory (excluding mild asthma in Part 2) or renal function, diabetes mellitus, coronary heart disease, cancer, or history of any psychotic mental illness
* Respiratory tract infection within 4 weeks before the screening visit
* History of surgery or medical intervention, or planned surgery or medical intervention
* Presence or history of severe adverse reaction to any drug, or sensitivity to components of the trial medication
* Use of a prescription or over-the-counter medicine, with the exception of acetaminophen (paracetamol), during the 7 days before the first dose of trial medication. For Part 2 only, inhaled short-acting ß2 agonists, and ICS (stable dose with at least 2 weeks documented use of ≥80% compliance before screening and Day -1) are permitted
* Participation in another clinical trial of a new chemical entity, new device, or a prescription medicine within the 3 months before dosing, or participation within 5 half-lives of receiving an experimental drug (whichever is longer)
* Presence or history of drug or alcohol abuse
* Evidence of drug abuse on urine testing, or a positive test for alcohol
* Current smoker; or ex-smokers who (a) gave up less than 1 year ago, or (b) who have a history of more than 10 pack-years
* Blood pressure and heart rate at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min.
* Loss of more than 400 mL blood, eg as a blood donor, or donation of blood products, during the 3 months before the trial
* Positive test for hepatitis B, hepatitis C, or HIV
* Possibility that the subject will not cooperate with the requirements of the protocol, including effective use of the DPI
* Additional exclusion criteria for Part 2:
* Life-threatening asthmatic episode in the past
* Asthmatic episode or respiratory tract infection requiring steroid treatment in the past 3 months
* Use of the following medicines within the specified time before screening:

  * Long-acting ß2 agonists; At any time before screening
  * Anti IgE therapy; 6 months
  * Inhaled corticosteroids (>500 µg per day of beclometasone dipropionate (BDP) or equivalent); 8 weeks
  * Oral or injectable steroids; 8 weeks
  * Intranasal or topical steroids; 4 weeks
  * Leukotriene antagonists; 2 weeks
  * Xanthines (excluding caffeine), anticholinergics, cromoglycates; 1 week

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of the safety and tolerability of single doses of VR942 in healthy subjects and repeated doses of VR942 in mild asthmatics | 28 days
  o Vital signs, physical examinations, any AEs or adverse device effects, laboratory tests, spirometry, and ECG variables

SECONDARY OUTCOMES:
The pharmacodynamics of repeat doses of VR942 in mild asthmatics | 28 days
  o Change in biomarker levels
The pharmacokinetic profile of single (Part 1) and repeated doses (part 2) of VR942 (time frame 4 and 14 days for Part 1 & 2 respectively): | 4 and 14 days for Part 1 and 2 respectively
  Part 1:
  Cmax, tmax, t½, AUC0-t, AUC0-∞ and Kel
  Part 2:
  Cmax, tmax, and AUC0-τ (post-dose on Day 1) Ctrough on Days 2, 9 and 10 Cmax, tmax, t½, AUC0-t, AUC0-τ, Kel (post-dose on Day 10) Accumulation ratio Racc (Cmax on Day 10/Cmax on Day 1), (AUC0-τ on Day 10/AUC0-τ on Day 1) and (Cmin on Day 10/Cmin on Day 2)
The number of used blisters and inhalers that do not meet the performance characteristics of the device intended by the manufacturer | 28 days
  o Examination of a sample of used blisters and inhalers will be conducted

CONTACTS AND LOCATIONS:
Locations (1):
- Vectura Study Site, London, United Kingdom

REFERENCES:
- [Derived] Burgess G, Boyce M, Jones M, Larsson L, Main MJ, Morgan F, Phillips P, Scrimgeour A, Strimenopoulou F, Vajjah P, Zamacona M, Palframan R. Randomized study of the safety and pharmacodynamics of inhaled interleukin-13 monoclonal antibody fragment VR942. EBioMedicine. 2018 Sep;35:67-75. doi: 10.1016/j.ebiom.2018.07.035. Epub 2018 Aug 23. PMID 30146344